CLINICAL TRIAL: NCT06740487
Title: Advanced Wireless Augmented Reality-Enhanced Exposure Therapy for Posttraumatic Stress Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arash Javanbakht, Director of Stress, Trauma, and Anxiety Research Clinic (STARC), Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUSC IRB#: Pro00135785; HT9425-24-1-0358 (Other Grant/Funding Number: U.S. Department of Defense)
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics; Elements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Exposure Therapy (ET) Treatment (Active Comparator): The active comparator group receives traditional prolonged exposure therapy alone, delivered in 60 minute sessions over 10 days across 5-10 weeks (sessions to occur 2-3x/week, with weekends off). Participants in both groups will be advised to continue in vivo exposure to real life situations (grocery shopping, going out, going to gatherings, etc.) in-between the sessions.
  Interventions: Behavioral: Traditional Exposure Therapy (ET) Treatment
- Traditional Exposure Therapy (ET) Treatment with addition of Augmented Reality (AR) Component (Experimental): Participants in the experimental group will begin with 10 60-minute sessions of in person ARET treatment across 5-10 weeks (sessions to occur 2-3x/week, with weekends off). This will involve wearing augmented reality (AR) goggles during exposure therapy to AR scenarios. At session 10, those with PCL score reduction of at least 12 points and a PCL score of below 33 (accepted diagnostic cut-off), will end treatment. Those who do not meet these criteria will continue with 10 sessions of 60-minute PE treatment across 5-10 weeks (sessions to occur 2-3x/week, with weekends off). Participants in both groups will be advised to continue in vivo exposure to real life situations (grocery shopping, going out, going to gatherings, etc.) in-between the sessions.
  Interventions: Behavioral: Stepwise Augmented Reality (AR) Component with Traditional Exposure Treatment for Nonresponders

INTERVENTIONS:
Behavioral: Traditional Exposure Therapy (ET) Treatment — Traditional exposure therapy (ET) includes the following components: (a) psychological education about trauma (sessions 1 and 2), (b) repeated in vivo exposure to trauma-related stimuli (in vivo exercises are assigned as homework during sessions 3 through 9), (c) repeated, prolonged, imaginal exposure to traumatic memories (imaginal exposure is implemented during sessions 3 - 9; patients listen to session audiotapes for homework between sessions), and (d) relapse prevention strategies and further treatment planning (session 10).
  Arms: Traditional Exposure Therapy (ET) Treatment
Behavioral: Stepwise Augmented Reality (AR) Component with Traditional Exposure Treatment for Nonresponders — The Augmented Reality Exposure Therapy component includes the following: (a) 60-minute sessions dedicated to augmented reality exposure therapy (ARET; sessions 1-10), (b) repeated in vivo exposure to trauma-related stimuli (in vivo exercises are assigned as homework during sessions 3 through 9), and (c) relapse prevention strategies and further treatment planning (session 10). During ARET, the clinician guides participant, who is wearing augmented reality (AR) goggles, through preset scenarios during which characters mingle with each other (e.g., grocery store, social gathering), as well as custom scenarios where participant can interact with the character. Those who do not respond to treatment (i.e., responders defined as PCL score reduction of at least 12 points and final PCL score below 33) will then subsequently participate in 10 60-minute sessions of traditional exposure therapy (ET) identical to procedures described for the traditional ET arm.
  Arms: Traditional Exposure Therapy (ET) Treatment with addition of Augmented Reality (AR) Component

SUMMARY:
The goal of this trial is to test how augmented reality exposure therapy (ARET) may potentiate the effects of traditional exposure therapy administered to U.S. military personnel diagnosed with PTSD. 40 adult males and females over the age of 18 that have served, or are currently serving, in the U.S. military, with a current diagnosis of PTSD, will be recruited. Participants will be randomized into two groups: 20 participants will receive ARET + traditional ET, with the remaining 20 to receive traditional ET only. The main questions this trial aims to answer are:

* what are the different clinical and psychosocial functioning outcomes between veterans/active-duty personnel with PTSD who receive ARET + traditional ET versus traditional ET only
* what are the differences in acceptance and satisfaction of treatment, between ARET + traditional ET and the traditional ET-only group

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) affects 12-14% of military personnel exposed to combat or military sexual trauma. Exposure therapy (ET) is the core of effective treatments for PTSD. During ET, patients are gradually exposed to avoided situations until fear/avoidance diminish. Despite its centrality in treatment, dropout from ET is high. Furthermore, while ET allocates significant therapist time to imaginal exposure to trauma memories, it relies on patients to independently engage in in vivo exposure to real-life situations they avoid (e.g., a crowded room or a grocery store). This limits patients' success in key exposure assignments, and importantly, their ability to return to civilian life functioning and work. Often, patients' symptoms improve, but social and occupational disability persists.

Augmented reality (AR) represents the newest wave of interactive human-computer technology, wherein virtual objects are mixed with physical reality. Instead of a completely synthetic environment (as with virtual reality; VR), AR simply adds to a patient's real physical context. As such, AR is less costly and easier to develop, and most importantly, is far more representative of the environment than VR, because AR IS the patient's environment, albeit with the addition of virtual feared stimuli.

To overcome ET limitations, researchers at the Stress, Trauma and Anxiety Research Clinic (STARC), in the Department of Psychiatry and Behavioral Neurosciences at Wayne State University, have created an AR technology that for the first time, allows the use of advanced AR technology for ET. This technology, called ExpandXR, is being used for treatment of first responders with PTSD. ExpandXR connects the clinician's computer to the AR headset via local area network (LAN) or Wi-Fi and provides a real-time 3D visual of the patient's surroundings on the therapist's computer. The clinician can see the position of the patient and the AR objects in a schematic of the room (not the real room), as well as the characters in patient's field of view. Simple clicks allow the clinician to control which virtual objects are present in the environment, as well as their behavior and movement. Stereo sound is delivered to the patient via speakers inside the headset. The software allows for recording of the number of augmented avatars in patient's field of view at any moment. Patients' subjective units of distress score (SUDS) can be directly entered into the software during the session.

ExpandXR includes 'scenarios' involving exposure to crowds in diverse social contexts. These scenarios have been designed by obtaining feedback from first responders, as well as the clinicians who work with them, while the technology has been developed in collaboration with experts with decades of experience in the gaming industry to ensure the realism needed for this application, and the highest possible overall quality of the product. The scenarios are scalable from very low on the fear hierarchy (e.g., two people talking to each other in a far corner of the room) to higher levels (e.g., a loud gathering with multiple groups of people, both in the patient's field of vision and behind them, with the sound of fireworks in the background). Current fixed scenarios include a gradually crowding party (which with some props could be transformed to a restaurant or bar), a gradually crowding grocery store, a bar/restaurant, a sports event, and office space. Some characters will have military fatigue on. Importantly, these scenarios include the normal life situations that are avoided by people with PTSD due to their trauma and are NOT recreations of the trauma memories. While engaged in a scenario, the patient, wearing the AR headset, can walk around, join groups, and listen to conversations. Some characters are interactive, walking towards the patient and addressing them directly. The clinician's desktop view livestreams the patient's position in space and their point of view (clinician can toggle between views). The exposure hierarchy intensity is easily increased or decreased by clicking arrows. The scenario can be paused and restarted. Sounds effect can be selected and adjusted for each patient. Patients' SUDS can be entered in real-time, and a data file with SUDS, timestamp and the level of exposure is exported at the end of the session. The software also has a library of near 100 diverse characters from which the clinician can choose and apply customized behaviors or interactions with a patient. The clinician can choose a character with specific physical characteristics, define their behavior, and type the content of their speech live. Of note, all these behaviors are normal life behaviors like walking, shaking head, nodding, tapping foot, smiling, looking surprised, etc. This aspect of the technology can be used for customized needs of each patient and their specific avoidances. The technology also allows automated conversations with AI driven characters, for practicing having a normal safe conversation with as stranger.

The technology has been well-received by first responders (a group with experiences relevant to military personnel) and pilot data suggest great success when used in treatment. Patients' initial resistance to ET seems to be an important limiting factor in acceptance of in vivo exposure. For the past several years, some findings from using ARET are that patients are more open to initiating treatment as they cognitively "know" the objects are not real. However, when engaged in the treatment, psychophysiological (SCR), behavioral, and subjective measures indicate that ARET elicits similar level of fear and arousal in response to virtual objects as to real feared objects.

This study will use a fine-tuned version of the above technology, which has been adjusted to specific civilian life needs of veterans and military personnel with PTSD, based on the feedback from national experts in military trauma, and veterans themselves.

Subject Recruitment:

40 adult males and females over the age of 18 that have served, or are currently serving, in the U.S. military, with a current diagnosis of PTSD, will be recruited. Subject recruitment will happen at the Ralph H. Johnson VA Healthcare System (RAJ VAHCS) in Charleston, South Carolina. Potential participants will be contacted by study staff when recruitment derives from the weekly PTSD clinic staff meetings at RAJ VAHCS. The investigators will also post flyers in the RHJ VAHCS, Charleston, and Savannah communities. Potential participants who respond to flyers, or who are referred by other providers, will be directed to the study coordinator where they will review informed consent and have all questions answered. If for any reason the study coordinator and patient cannot meet face-to-face, participants may be contacted via telephone to discuss study parameters. The investigators will also list this study among those listed in our consortium institution's (Medical University of South Carolina) "scresearch.org" web page. Also, primary care and mental health providers of veterans for whom PTSD is suspected may also refer to the study. For individuals that do not meet study inclusion criteria, the study staff will assist with coordinating appropriate care outside of the study.

Treatment will take place at the Ralph H. Johnson VA Healthcare System (RAJ VAHCS) in Charleston, South Carolina. This study involves administering a full course of integrated ARET + ET treatment for PTSD to 20 patients and administering ET treatment for PTSD alone to 20 others. Participants will be randomly assigned to receive ARET + ET or ET alone. Both groups will receive 10 60-minute sessions. Participants in the ARET + ET group will begin with 10 sessions of in person ARET treatment. At session 10, those whose PCL score has reduced at least 12 points from baseline and whose score is less than 33 (diagnostic cutoff), will end treatment. Those who do not meet these two criteria will continue with 10 sessions of 60-minute PE treatment. This stepwise approach, especially in the context of this feasibility clinical trial, will a) inform stepped care practice, b) assess whether in some or all patients ARET can serve as a lower burden, first line intervention, and c) reduce the time commitment in each session, instead of longer ARET + PE in one session. ARET sessions will be in person. Consistent with VA PTSD clinic standards, for both groups, PE treatment sessions will be offered in person or via home telehealth in both conditions.

Participants in the ARET group will be fitted with the AR goggles, and the clinician will see the patient's point of view on a desktop computer. The clinician will explain each of the preset scenarios to the patient (e.g., crowded gathering, grocery store, restaurant, bar, office space), and then start with the scenario that patient indicates they find the easiest. The hierarchies of these scenarios are preset and the same for all participants, which mostly involves addition of more characters. At each level, when the patient's SUDS score is 4 or below and the patient gives the go-ahead, the scenario will be increased to the next level. Patients are assured that they will not be surprised, and nothing will happen without their approval. Participants will also be told that they can stop/pause the scenarios at any time. When the first scenario is completed and the patient has SUDS of 4 or below at the highest level of hierarchy exposure, the clinician will leave the room, to allow a sense of control, which is very important for autonomy in real life. Clinician will still be available via intercom.

Throughout the sessions, when each scenario is completed, the patients will move on to another scenario, until they have successfully completed all the scenarios, or have decided to not continue any specific scenario. After that, the clinician will use characters from the character library, and create interactive situations based on specific needs of each patient. Therapy will be conducted based on the principles of conventional exposure therapy. During the exposure, the provider can be in the same room, or a different room in the clinic, but will still be connected to the patient through voice. At any time, if the level of distress due to exposure is determined to be too high, both the patient and the provider can pause or terminate the exposure.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female over the age of 18 that has served, or is currently serving, in the military.
* Current diagnosis of PTSD as determined by a Clinician Administered PTSD Scale for DSM-5 (CAPS-5) clinical interview.

Exclusion Criteria:

* Active psychosis or dementia at screening.
* Suicidal ideation with clear intent.
* Concurrent enrollment in another clinical trial for PTSD or depression.
* Substance use disorders
* Visual impairments not allowing use of augmented reality. Visual impairments that are corrected with contact lens visual aid are not considered exclusionary as contacts can be worn under the AR headset. For patients with vision impairment that cannot wear contacts, a diopter value no stronger than -2.00 is acceptable.

Exclusion criteria are limited to those factors that would negatively impact the validity of the study findings, or place participants at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale-5 Revised (CAPS-5 R) - past week | Change in score from baseline to post treatment (immediately following the 10th exposure therapy session).
  The CAPS-5 R is a 30-item structured interview conducted by a clinician with a patient, to assess for presence of PTSD and/or severity of PTSD symptoms, according to the DSM-5 criteria (prior text generated with help of AI). For each item, the clinician asks the patient the frequency with which they've had a specific problem in the past month, in addition to more specific questions depending on the problem being explored.
Clinician Administered PTSD Scale-5 Revised (CAPS-5 R) - past week | Change in score from baseline to post treatment, 3-months after last exposure therapy session
  The CAPS-5 R is a 30-item structured interview conducted by a clinician with a patient, to assess for presence of PTSD and/or severity of PTSD symptoms, according to the DSM-5 criteria (prior text generated with help of AI). For each item, the clinician asks the patient the frequency with which they've had a specific problem in the past month, in addition to more specific questions depending on the problem being explored.
Clinician Administered PTSD Scale-5 Revised (CAPS-5 R) - past week | Change in score from baseline to post treatment, 6-months after last exposure therapy session
  The CAPS-5 R is a 30-item structured interview conducted by a clinician with a patient, to assess for presence of PTSD and/or severity of PTSD symptoms, according to the DSM-5 criteria (prior text generated with help of AI). For each item, the clinician asks the patient the frequency with which they've had a specific problem in the past month, in addition to more specific questions depending on the problem being explored.
Liebowitz Social Anxiety Scale (LSAS-SR) | Change in score from baseline to post treatment (immediately following the 10th exposure therapy session).
  The LSAS-SR is a 24-item structured interview conducted by a clinician with a patient, that assesses for presence of social anxiety disorder. Each item asks two questions about the particular item. Respondents rate the first question of the item on a 4-point Likert scale ranging from 0 ("None") to 3 ("Severe"), indicating how anxious or fearful they feel in a specific situation. Respondents rate the second question of the item on a 4-point Likert scale ranging from 0 ("Never") to 3 ("Usually") indicating how often they avoid a specific situation.
Liebowitz Social Anxiety Scale (LSAS-SR) | Change in score from baseline to post treatment, 3-months after last exposure therapy session
  The LSAS-SR is a 24-item structured interview conducted by a clinician with a patient, that assesses for presence of social anxiety disorder. Each item asks two questions about the particular item. Respondents rate the first question of the item on a 4-point Likert scale ranging from 0 ("None") to 3 ("Severe"), indicating how anxious or fearful they feel in a specific situation. Respondents rate the second question of the item on a 4-point Likert scale ranging from 0 ("Never") to 3 ("Usually") indicating how often they avoid a specific situation.
Liebowitz Social Anxiety Scale (LSAS-SR) | Change in score from baseline to post treatment, 6-months after last exposure therapy session
  The LSAS-SR is a 24-item structured interview conducted by a clinician with a patient, that assesses for presence of social anxiety disorder. Each item asks two questions about the particular item. Respondents rate the first question of the item on a 4-point Likert scale ranging from 0 ("None") to 3 ("Severe"), indicating how anxious or fearful they feel in a specific situation. Respondents rate the second question of the item on a 4-point Likert scale ranging from 0 ("Never") to 3 ("Usually") indicating how often they avoid a specific situation.
PTSD Checklist (PCL5) - past week | Change in score from baseline to post treatment (immediately following the 10th exposure therapy session).
  The PCL-5_Past Week is a 20-item structured interview conducted by a clinician with a patient, that assesses presence and severity of PTSD symptoms related to a very stressful experience. Respondents rate each item on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Extremely"), indicating how much they have been bothered by each symptom in the past week.
PTSD Checklist (PCL5) - past week | Change in score from baseline to post treatment, 3-months after last exposure therapy session
  The PCL-5_Past Week is a 20-item structured interview conducted by a clinician with a patient, that assesses presence and severity of PTSD symptoms related to a very stressful experience. Respondents rate each item on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Extremely"), indicating how much they have been bothered by each symptom in the past week.
PTSD Checklist (PCL5) - past week | Change in score from baseline to post treatment, 6-months after last exposure therapy session
  The PCL-5_Past Week is a 20-item structured interview conducted by a clinician with a patient, that assesses presence and severity of PTSD symptoms related to a very stressful experience. Respondents rate each item on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Extremely"), indicating how much they have been bothered by each symptom in the past week.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale 5 Revised (CAPS-5 R) | Change in score from baseline to post-treatment (Week 20; immediately following completion of the 20th session for participants who complete ARET+PE)
  The CAPS-5 R is a 30-item structured interview conducted by a clinician with a patient, to assess for presence of PTSD and/or severity of PTSD symptoms, according to the DSM-5 criteria (prior text generated with help of AI). For each item, the clinician asks the patient the frequency with which they've had a specific problem in the past month, in addition to more specific questions depending on the problem being explored.
Liebowitz Social Anxiety Scale (LSAS-SR) | Change in score from baseline to post-treatment (Week 20; immediately following completion of the 20th session for participants who complete ARET+PE)
  The LSAS-SR is a 24-item structured interview conducted by a clinician with a patient, that assesses for presence of social anxiety disorder. Each item asks two questions about the particular item. Respondents rate the first question of the item on a 4-point Likert scale ranging from 0 ("None") to 3 ("Severe"), indicating how anxious or fearful they feel in a specific situation. Respondents rate the second question of the item on a 4-point Likert scale ranging from 0 ("Never") to 3 ("Usually") indicating how often they avoid a specific situation.
PTSD Checklist (PCL5) | Change in score from baseline to post-treatment (Week 20; immediately following completion of the 20th session for participants who complete ARET+PE)
  The PCL-5_Past Week is a 20-item structured interview conducted by a clinician with a patient, that assesses presence and severity of PTSD symptoms related to a very stressful experience. Respondents rate each item on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Extremely"), indicating how much they have been bothered by each symptom in the past week.
Social Functioning Questionnaire (AI generated) | Change in score from baseline to post treatment (immediately following the 10th exposure therapy session).
  The Social Functioning Questionnaire (AI generated) is a 10-item self-report questionnaire that assesses presence of social dysfunction across various situations of daily living. Respondents rate each item on a 5-point Likert scale ranging from 0 ("Never") to 5 ("Always"), indicating how much they have been bothered by the situation in the past week.
Social Functioning Questionnaire (AI generated) | Change in score from baseline to post-treatment (Week 20; immediately following completion of the 20th session for participants who complete ARET+PE)
  The Social Functioning Questionnaire (AI generated) is a 10-item self-report questionnaire that assesses presence of social dysfunction across various situations of daily living. Respondents rate each item on a 5-point Likert scale ranging from 0 ("Never") to 5 ("Always"), indicating how much they have been bothered by the situation in the past week.
Social Functioning Questionnaire (AI generated) | Change in score from baseline to post treatment, 3-months after last exposure therapy session
  The Social Functioning Questionnaire (AI generated) is a 10-item self-report questionnaire that assesses presence of social dysfunction across various situations of daily living. Respondents rate each item on a 5-point Likert scale ranging from 0 ("Never") to 5 ("Always"), indicating how much they have been bothered by the situation in the past week.
Social Functioning Questionnaire (AI generated) | Change in score from baseline to post treatment, 6-months after last exposure therapy session
  The Social Functioning Questionnaire (AI generated) is a 10-item self-report questionnaire that assesses presence of social dysfunction across various situations of daily living. Respondents rate each item on a 5-point Likert scale ranging from 0 ("Never") to 5 ("Always"), indicating how much they have been bothered by the situation in the past week.
Post-Traumatic Avoidance Behavior Questionnaire (PABQ) | Change in score from baseline to post treatment (immediately following the 10th exposure therapy session).
  The PABQ is a 25-item self-report questionnaire that measures avoidance behavior related to a traumatic experience. Respondents rate each item on a 4-point Likert scale ranging from 0 ("(Almost) Never"), to 4 "(Almost) Always"), indicating how often they engaged in certain behaviors over the past 4 weeks.
Post-Traumatic Avoidance Behavior Questionnaire (PABQ) | Change in score from baseline to post-treatment (Week 20; immediately following completion of the 20th session for participants who complete ARET+PE)
  The PABQ is a 25-item self-report questionnaire that measures avoidance behavior related to a traumatic experience. Respondents rate each item on a 4-point Likert scale ranging from 0 ("(Almost) Never"), to 4 "(Almost) Always"), indicating how often they engaged in certain behaviors over the past 4 weeks.
Post-Traumatic Avoidance Behavior Questionnaire (PABQ) | Change in score from baseline to post treatment, 3-months after last exposure therapy session
  The PABQ is a 25-item self-report questionnaire that measures avoidance behavior related to a traumatic experience. Respondents rate each item on a 4-point Likert scale ranging from 0 ("(Almost) Never"), to 4 "(Almost) Always"), indicating how often they engaged in certain behaviors over the past 4 weeks.
Post-Traumatic Avoidance Behavior Questionnaire (PABQ) | Change in score from baseline to post treatment, 6-months after last exposure therapy session
  The PABQ is a 25-item self-report questionnaire that measures avoidance behavior related to a traumatic experience. Respondents rate each item on a 4-point Likert scale ranging from 0 ("(Almost) Never"), to 4 "(Almost) Always"), indicating how often they engaged in certain behaviors over the past 4 weeks.
UCLA-Loneliness Scale (short form) | Change in score from baseline to post treatment (immediately following the 10th exposure therapy session).
  The UCLA-Loneliness scale (short form) is a 3-item self-report questionnaire that assesses the frequency of feelings of loneliness. Respondents rate each item on a 3-point Likert scale ranging from 1 ("Hardly ever") to 3 ("Often").
UCLA-Loneliness Scale (short form) | Change in score from baseline to post-treatment (Week 20; immediately following completion of the 20th session for participants who complete ARET+PE)
  The UCLA-Loneliness scale (short form) is a 3-item self-report questionnaire that assesses the frequency of feelings of loneliness. Respondents rate each item on a 3-point Likert scale ranging from 1 ("Hardly ever") to 3 ("Often").
UCLA-Loneliness Scale (short form) | Change in score from baseline to post treatment, 3-months after last exposure therapy session
  The UCLA-Loneliness scale (short form) is a 3-item self-report questionnaire that assesses the frequency of feelings of loneliness. Respondents rate each item on a 3-point Likert scale ranging from 1 ("Hardly ever") to 3 ("Often").
UCLA-Loneliness Scale (short form) | Change in score from baseline to post treatment, 6-months after last exposure therapy session
  The UCLA-Loneliness scale (short form) is a 3-item self-report questionnaire that assesses the frequency of feelings of loneliness. Respondents rate each item on a 3-point Likert scale ranging from 1 ("Hardly ever") to 3 ("Often").
Credibility Expectancy Questionnaire | Change in score from baseline to post treatment (immediately following the 10th exposure therapy session).
  The Credibility Expectancy Questionnaire is a 6-item self-report questionnaire that assesses how much a respondent believes the treatment they're receiving will help improve their lifestyle/functioning. Respondents rate each item on a 9-point Likert scale ranging from 1 to 9, with 1 being the low score and 9 being the highest. Total score is calculated by adding all items together. Higher scores are indicative of greater expectancy in treatment credibility and efficacy.
Credibility Expectancy Questionnaire | Change in score from baseline to post-treatment (Week 20; immediately following completion of the 20th session for participants who complete ARET+PE)
  The Credibility Expectancy Questionnaire is a 6-item self-report questionnaire that assesses how much a respondent believes the treatment they're receiving will help improve their lifestyle/functioning. Respondents rate each item on a 9-point Likert scale ranging from 1 to 9, with 1 being the low score and 9 being the highest. Total score is calculated by adding all items together. Higher scores are indicative of greater expectancy in treatment credibility and efficacy.
Credibility Expectancy Questionnaire | Change in score from baseline to post treatment, 3-months after last exposure therapy session
  The Credibility Expectancy Questionnaire is a 6-item self-report questionnaire that assesses how much a respondent believes the treatment they're receiving will help improve their lifestyle/functioning. Respondents rate each item on a 9-point Likert scale ranging from 1 to 9, with 1 being the low score and 9 being the highest. Total score is calculated by adding all items together. Higher scores are indicative of greater expectancy in treatment credibility and efficacy.
Credibility Expectancy Questionnaire | Change in score from baseline to post treatment, 6-months after last exposure therapy session
  The Credibility Expectancy Questionnaire is a 6-item self-report questionnaire that assesses how much a respondent believes the treatment they're receiving will help improve their lifestyle/functioning. Respondents rate each item on a 9-point Likert scale ranging from 1 to 9, with 1 being the low score and 9 being the highest. Total score is calculated by adding all items together. Higher scores are indicative of greater expectancy in treatment credibility and efficacy.
Patient Health Questionnaire-9 (PHQ-9) | Change in score from baseline to post treatment (immediately following the 10th exposure therapy session).
  The PHQ-9 is a 9-item self-report questionnaire that assesses severity of depression symptoms over the past two weeks. Respondents rate each item on a 4-point Likert scale ranging from 0 ("Not at all") to 4 ("Nearly every day"), indicating how much they have been bothered by each symptom over the past two weeks.
Patient Health Questionnaire-9 (PHQ-9) | Change in score from baseline to post-treatment (Week 20; immediately following completion of the 20th session for participants who complete ARET+PE)
  The PHQ-9 is a 9-item self-report questionnaire that assesses severity of depression symptoms over the past two weeks. Respondents rate each item on a 4-point Likert scale ranging from 0 ("Not at all") to 4 ("Nearly every day"), indicating how much they have been bothered by each symptom over the past two weeks.
Patient Health Questionnaire-9 (PHQ-9) | Change in score from baseline to post treatment, 3-months after last exposure therapy session
  The PHQ-9 is a 9-item self-report questionnaire that assesses severity of depression symptoms over the past two weeks. Respondents rate each item on a 4-point Likert scale ranging from 0 ("Not at all") to 4 ("Nearly every day"), indicating how much they have been bothered by each symptom over the past two weeks.
Patient Health Questionnaire-9 (PHQ-9) | Change in score from baseline to post treatment, 6-months after last exposure therapy session
  The PHQ-9 is a 9-item self-report questionnaire that assesses severity of depression symptoms over the past two weeks. Respondents rate each item on a 4-point Likert scale ranging from 0 ("Not at all") to 4 ("Nearly every day"), indicating how much they have been bothered by each symptom over the past two weeks.
Satisfaction with Social Roles and Activities - Short Form 8a (PROMIS) | Change in score from baseline to post-treatment (immediately following the 10th exposure therapy session)
  The PROMIS Satisfaction with Social Roles and Activities - Short Form 8a is an 8-item self-report questionnaire that assesses an individual's perceived satisfaction with their ability to perform and participate in usual social roles and activities (e.g., work, family responsibilities, and social interactions). Respondents rate each item on a 5-point Likert scale, reflecting the extent of their satisfaction over the specified time period, with higher scores indicating greater satisfaction with social functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Acierno, PhD, Principal Investigator — Ralph H. Johnson VA Health Care System
Locations (1):
- Ralph H. Johnson VA Health Care System, Charleston, South Carolina, United States

REFERENCES:
- [Background] Chu JA. Posttraumatic stress disorder: Beyond DSM-IV. Am J Psychiatry. 2010 Jun;167(6):615-7. doi: 10.1176/appi.ajp.2010.10030310. No abstract available. PMID 20516157
- [Background] Keane TM, Wolfe J. Comorbidity in post-traumatic stress disorder: An analysis of community and clinical studies. Journal of Applied Social Psychology. 1990;20(21, Pt 1):1776-1788. doi:10.1111/j.1559-1816.1990.tb01511.x
- [Background] Kulka RA, Schlenger WE, Fairbank JA, et al. Trauma and the Vietnam war generation: Report of findings from the National Vietnam Veterans Readjustment Study. Trauma and the Vietnam war generation: Report of findings from the National Vietnam Veterans Readjustment Study. Brunner/Mazel; 1990:xxix, 322-xxix, 322.
- [Background] Dohrenwend BP, Turner JB, Turse NA, Adams BG, Koenen KC, Marshall R. The psychological risks of Vietnam for U.S. veterans: a revisit with new data and methods. Science. 2006 Aug 18;313(5789):979-82. doi: 10.1126/science.1128944. PMID 16917066
- [Background] Fulton JJ, Calhoun PS, Wagner HR, Schry AR, Hair LP, Feeling N, Elbogen E, Beckham JC. The prevalence of posttraumatic stress disorder in Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans: a meta-analysis. J Anxiety Disord. 2015 Apr;31:98-107. doi: 10.1016/j.janxdis.2015.02.003. Epub 2015 Feb 19. PMID 25768399
- [Background] Frueh BC, Elhai JD, Grubaugh AL, Monnier J, Kashdan TB, Sauvageot JA, Hamner MB, Burkett BG, Arana GW. Documented combat exposure of US veterans seeking treatment for combat-related post-traumatic stress disorder. Br J Psychiatry. 2005 Jun;186:467-72; discussion 473-5. doi: 10.1192/bjp.186.6.467. PMID 15928355
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Hoge CW, Auchterlonie JL, Milliken CS. Mental health problems, use of mental health services, and attrition from military service after returning from deployment to Iraq or Afghanistan. JAMA. 2006 Mar 1;295(9):1023-32. doi: 10.1001/jama.295.9.1023. PMID 16507803
- [Background] Foa EB, Hembree EA, Rothbaum BO. Prolonged exposure therapy for PTSD: Emotional processing of traumatic experiences: Therapist guide. Prolonged exposure therapy for PTSD: Emotional processing of traumatic experiences: Therapist guide. Oxford University Press; 2007:viii, 146-viii, 146.
- [Background] Kehle-Forbes SM, Meis LA, Spoont MR, Polusny MA. Treatment initiation and dropout from prolonged exposure and cognitive processing therapy in a VA outpatient clinic. Psychol Trauma. 2016 Jan;8(1):107-114. doi: 10.1037/tra0000065. Epub 2015 Jun 29. PMID 26121175
- [Background] Bouton ME, Bolles RC. Contextual control of the extinction of conditioned fear. Learning and Motivation. 1979/11/01/ 1979;10(4):445-466. doi:https://doi.org/10.1016/0023-9690(79)90057-2
- [Background] Javanbakht A, Madaboosi S, Grasser LR. Real-life contextualization of exposure therapy using augmented reality: A pilot clinical trial of a novel treatment method. Ann Clin Psychiatry. 2021 Nov;33(4):220-231. doi: 10.12788/acp.0042. PMID 34672925
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509